CLINICAL TRIAL: NCT00576680
Title: Phase I/II Study of RAD001 in Combination With Temozolomide in Patients With Advanced Pancreatic Neuroendocrine Tumors
Brief Title: RAD001 and Temozolomide in Patients With Advanced Pancreatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Novartis (Industry); Schering-Plough (Industry)
Responsible Party: Principal Investigator, Jennifer Chan, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-325
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Pancreatic Neuroendocrine Tumor
Keywords: RAD001; temozolomide
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Everolimus; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide with RAD001 (Experimental)
  Interventions: Drug: RAD001; Drug: Temozolomide

INTERVENTIONS:
Drug: RAD001 — Given orally once a day
Drug: Temozolomide — Taken orally once a day for one week followed by a one-week break period
  Other Names: Temodar

SUMMARY:
This research study will test the safety of RAD001 in combination with temozolomide.

DETAILED DESCRIPTION:
* Participants will take RAD001 by mouth daily. They will also take temozolomide by mouth daily for one week, followed by a one-week break period. This one-week on/one week off schedule for temozolomide will continue for the duration of the treatment.
* After the first month of treatment, there will be a 7-day observation period during which no study medication will be taken to observe for any side effects.
* During all treatment cycles (1 cycle is 28 days in length) participants will have a physical exam and will be asked questions about their general health and specific questions about any problems they may be experiencing. Initially, participants will come in every other week. At each of these visits, blood work will be taken to monitor the participants health.
* After every 2 months of treatment, participants will have a CT scan or MRI done to see how the medication is working.

ELIGIBILITY:
Inclusion Criteria:

* Locally unresectable or metastatic pancreatic neuroendocrine tumor
* Radiologic, operative, or pathology reports should document a pancreatic location of tumor
* Patients must have confirmed low-grade or intermediate-grade neuroendocrine carcinoma
* Patients must have at least one measurable site of disease according to RECIST criteria that has not been preciously irradiated
* 18 years of age or older
* Minimum of two weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy
* Prior treatment with chemotherapy is allowed, with the exception of prior treatment with temozolomide or dacarbazine
* No Prior therapy with RAD001 or any other mTOR inhibitor
* ECOG Performance status 0,1 or 2
* Life expectancy 12 weeks or more
* Adequate bone marrow, liver and renal function as outlined in the protocol
* Negative serum pregnancy test
* Fasting serum cholesterol as outlined in protocol

Exclusion Criteria:

* Prior treatment with any investigational drug within the preceding 4 weeks
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinoma of the skin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Women who are pregnant or breast feeding
* Patients who have received prior treatment with an mTOR inhibitor or temozolomide
* Patients with known hypersensitivity to RAD001 or other rapamycins or to its excipients
* History of noncompliance to medical regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-05; Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Chan, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Temozolomide and Everolimus: Temozolomide was administered to all patients at a starting dose of 150 mg/m2 on days 1 to 7 and days 15 to 21 of a 28-day cycle. Everolimus was administered together with temozolomide in 2 dose cohorts: 1) 5 mg daily and 2) 10 mg daily.
Period: Overall Study
Arm/Group | Temozolomide and Everolimus
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide and Everolimus
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 53 [28 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: To determine the objective response rate by RECIST criteria of RAD001 in combination with temozolomide in patients with advanced pancreatic neuroendocrine tumors. Partial response (PR) by these criteria is defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Progressive disease (PD) is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions. Stable Disease (SD) is defined as neither sufficient decrease to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide and Everolimus
Number analyzed (Participants) | 40
Participants | 16

2. Secondary Outcome: Progression-free Survival
Description: To determine progression-free survival when RAD001 is given in combination with temozolomide in patients with advanced pancreatic neuroendocrine tumors. Progression-free survival is defined as time from start of therapy until disease progression, as defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions, or death.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide and Everolimus
Number analyzed (Participants) | 43
months | 15.4 [9.4 to 20.4]

3. Secondary Outcome: To Determine the Safety and Tolerability of This Drug Combination.
Description: To determine the safety and tolerability of RAD001 when given in combination with temozolomide in patients with advanced pancreatic neuroendocrine tumors.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide and Everolimus
Number analyzed (Participants) | 43
Participants
  Grade 3 or 4 Lymphopenia | 19
  Grade 3 or 4 thrombocytopenia | 7
  Grade 3 or 4 mucositis | 1
  Grade 3 or 4 hyperglycemia | 8
  Grade 3 or 4 AST Increase | 4
  Grade 3 or 4 Leukocyte decrease | 7

ADVERSE EVENTS:
Time Frame: Participants were followed for development of adverse events for the entire duration while receiving treatment and for 30 days following their last dose of study treatment. Patients in this trial received a median of 8.5 four-week treatment cycles (range, 1-28). Each participant was followed for adverse events for 30 days following his or her last dose of study treatment.
Description: All-grade adverse events possible or definitely related to treatment are reported.
Arm/Group | Temozolomide and Everolimus
All-Cause Mortality (participants affected / at risk) | 2/43
Serious Adverse Events (participants affected / at risk) | 15/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide and Everolimus (N=43)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
neutropenia (Blood and lymphatic system disorders) | 2 (2)
hypocalcemia (Investigations) | 1 (1)
creatinine (Renal and urinary disorders) | 0 (0)
hypophosphatemia (Investigations) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
lymphopenia (Blood and lymphatic system disorders) | 8 (10)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide and Everolimus (N=43)
Fatigue (General disorders) | 33
Nausea (Gastrointestinal disorders) | 33
Mucositis (Gastrointestinal disorders) | 27
Hyperglycemia (Endocrine disorders) | 31
Hypercholesterolemia (General disorders) | 18
Lymphocytopenia (Blood and lymphatic system disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT00576680/Prot_SAP_000.pdf